CLINICAL TRIAL: NCT00890838
Title: Preoperative Intravenous Omega 3 Fatty Acids Administration in Valvular Surgery Patients: A Prospective, Randomized, Open-label, Comparative Clinical Trial
Brief Title: Preoperative Intravenous Omega 3 Fatty Acids Administration in Valvular Surgery Patients
Acronym: IVFO-Valvular
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nizam's Institute of Medical Sciences University, India (Other)
Responsible Party: Principal Investigator, Dr. R. Gopinath, Professor, Nizam's Institute of Medical Sciences University, India
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NIMS/2008/Omegaven/Surgery/02
Record Dates: First submitted 2009-04-28; First posted 2009-04-30 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-10

CONDITIONS: Valvular Surgery; Inflammation
Keywords: IVFO; Inflammation; Valvular surgery; Inflammatory status; Infectious complications
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omegaven (Active Comparator): will receive IV Omega 3 fatty acids (Omegaven®) for 3 days preoperatively
  Interventions: Dietary Supplement: Omegaven-IV FO
- Without Omegaven (No Intervention): will not receive IV Omega 3 fatty acids (Omegaven®) for 3 days preoperativel

INTERVENTIONS:
Dietary Supplement: Omegaven-IV FO — will receive IV Omega 3 fatty acids (Omegaven®) for 3 pre operative days
  Arms: Omegaven

SUMMARY:
The perioperative administration of n-3 fatty acids has been shown to lead to favorable effects on outcome in patients with severe surgical interventions by lowering the magnitude of inflammatory response and by modulating the immune response. To the investigators' knowledge, no study with preoperative administration of intravenous (IV) omega 3 fatty acids as a part of total parenteral nutrition (TPN) or monotherapy with it to demonstrate its effects on inflammatory and immune response has been conducted. So, this study has been planned to judge the inflammatory response of preoperative monotherapy with IV omega 3 fatty acids in elderly patients undergoing valvular surgery considering the hyperinflammation associated with this type of surgery in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female patients undergoing valvular surgeries
2. Age 18-50 years
3. The patients who give written informed consent

Exclusion Criteria:

1. Refusal to participate in the study
2. Allergy to any of the constituents of nutritional products
3. HIV positive patients, patients with primary diagnosis of hypertriglyceridemia, patients on long term steroid therapy and cycloxygenase inhibitors (more than 3 months)
4. Severe cardiac disease, hepatic disorders (total bilirubin > 1.5 times the upper limit of normal), psychiatric disorders likely to affect compliance, severe hemorrhagic disorders, stroke, embolism
5. Uncontrolled severe renal failure (Serum creatinine > 2 mg/dL) without dialysis/hemofiltration
6. Pregnant or nursing women
7. Participation in any other clinical trial within the last 2 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-04; Primary Completion 2010-04 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
IL-6, 8, 10, HS-CRP | 5 days

SECONDARY OUTCOMES:
Infectious complications | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Dr R Gopinath, Principal Investigator — Professor and Head, Department of ANesthesia and critical care
Locations (1):
- NIzam's Institute of Medical Sciences, Hyderabad, Andhra Pradesh, India